CLINICAL TRIAL: NCT07334275
Title: Pilot Study for the Detection of Minimal Residual Disease Post-prostatectomy and Early Disease Recurrence in Circulating Tumor DNA to Guide Future Adjuvant Therapy in High-risk Prostate Cancer Patients (MiRaDE)
Brief Title: Detection of Minimal Residual Disease Post-prostatectomy
Acronym: MiRaDE
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other); Canisius-Wilhelmina Hospital (Other); Maxima Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-18163
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Prostatectomy; Circulating tumor DNA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumor DNA (ctDNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-risk localized prostate cancer or high-risk locally advanced prostate cancer: Included patients will have:
  1. High-risk localized prostate cancer, with PSA level >20 ng/mL, Gleason score 8-10 (ISUP grade 4/5) at prostate biopsies, or iT3a (based on multi-parametric MRI of the prostate); or
  2. High-risk locally advanced prostate cancer, having any PSA level, any Gleason score/ISUP grade, iT3b-4 (based on multi-parametric MRI of the prostate) or iN1 (based on PSMA PET/CT imaging).

SUMMARY:
The clinical objective for this pilot study is to determine whether minimal residual disease (MRD) detection in high-risk prostate cancer, utilizing a custom-made prostate-specific circulating tumor DNA (ctDNA) panel, may lead to more optimal prediction of disease recurrence following radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 years or older;
* High-risk prostate cancer, defined as:

  1. High-risk localized prostate cancer, with PSA level >20 ng/mL, Gleason score 8-10 (ISUP grade 4/5) at prostate biopsies, or iT3a (based on multi-parametric MRI of the prostate); or
  2. High-risk locally advanced prostate cancer, having any PSA level, any Gleason score/ISUP grade, iT3b-4 (based on multi-parametric MRI of the prostate) or iN1 (based on PSMA PET/CT imaging);
* Scheduled for robot-assisted radical prostatectomy;
* Willingness to consent to both patient information sheets regarding tissue and liquid biobanking.

Exclusion Criteria:

* Relevant contra-indications that may limit clinical follow-up or blood collection, as assessed by the including physician.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-risk prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of high-risk prostate cancer patients in which ctDNA-detected minimal residual disease (MRD) exceeds 15% | From enrollment to 6 weeks postoperatively
  To determine the proportion of high-risk prostate cancer patients with ctDNA-detected minimal residual disease (MRD) at six weeks postoperatively
The relation between distant disease-free survival (DDFS) <12 months and minimal residual disease (MRD) positive patients | From enrollment to 12 months postoperatively
  To determine the risk of early relapse (radiological distant disease-free survival within twelve months following prostatectomy) in patients with and without ctDNA-detected minimal residual disease (MRD)

SECONDARY OUTCOMES:
The relation between distant disease-free survival (DDFS) and 12-week ctDNA-positive patients | From enrollment to 12 months postoperatively
  To determine the proportion of HR-PCa with ctDNA-detected early relapse at 12 weeks postoperatively
The relation between ctDNA% and distant disease-free survival (DDFS) | From enrollment to 12 months postoperatively
  To determine the preoperative ctDNA fractional abundance (ctDNA%) and the prognostic characteristics of ctDNA% related to early relapse and radiological disease-free survival
The relation between poor prognostic gene signature (TP53 and/or PTEN) and/or DNA damage repair alterations and distant disease-free survival (DDFS) | From enrollment to 12 months postoperatively
  To determine whether mutations in TP53, PTEN and DNA damage repair are associated with early distant metastasis-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Prosper Prostate Cancer Clinics, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided